CLINICAL TRIAL: NCT03830619
Title: Serum Exosomal Long Noncoding RNAs as Potential Biomarkers for Lung Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: WuhanUH2018
Record Dates: First submitted 2019-01-24; First posted 2019-02-05 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: exosomes；lncRNA； lung cancer；
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lung cancer patients
  Interventions: Diagnostic Test: collect samples
- normol volunteers
  Interventions: Diagnostic Test: collect samples

INTERVENTIONS:
Diagnostic Test: collect samples — collect serum samples and clinical features

SUMMARY:
The study is to investigate the sensitivity and specificity of serum exosome noncoding RNA as a biomarker for the diagnosis of lung cancer

DETAILED DESCRIPTION:
Conventional tumor markers for non-invasive diagnosis of Lung cancer (LC) exhibit insufficient sensitivity and specificity to facilitate detection of early lung cancer (ELC). The investigators aimed to identify ELC-specific exosomal lncRNA biomarkers that are highly sensitive and stable for the non-invasive diagnosis of ELC.Hence, in the present study, exosomes from the plasma of five healthy individuals and 30 LC patients and from culture media of four human bronchial epithelial cells and four cancer cells were isolated. Exosomal RNA profiling was performed using RNA sequencing to identify LC specific exosomal lncRNAs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are willing to sign the informed consent form;
* Normal subjects have no evidence of any disease;
* Lung cancer patients are 18 to 75 years old, diagnosed as lung cancer by histopathology or cytopathology

Exclusion Criteria:

* People are unwilling to sign the informed consent form;
* Patients with heart disease, rheumatic disease, allergic disease, COPD, pulmonary fibrosis, diabetes, thyroid disease, liver, kidney, brain disease and hematopoietic system disease;
* Pregnant or lactating women;
* Patients did not cooperate or participate in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as lung cancer by histopathology or cytopathology in union hospital.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The expression levels of serum exosome long non-coding RNA | the first day subjects are enrolled the outcome will be assessed；up to three years after the completion of the study
the expression levels of tumor biomarkers such as CEA, NSE, SCC, CYFR2A-1 | the first day subjects are enrolled the outcome will be assessed；up to three years after the completion of the study
the CT scans of the lung for the patients | the first day subjects are enrolled the outcome will be assessed；up to three years after the completion of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD now